CLINICAL TRIAL: NCT00519077
Title: Phase II Study of Skin Toxicity Dosing of IRESSA (Gefitinib) as Monotherapy in Recurrent and/or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Phase II Study of Skin Toxicity Dosing of IRESSA (Gefitinib) in Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13503A
Record Dates: First submitted 2007-08-17; First posted 2007-08-21 (Estimated); Results first posted 2013-11-21 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Head and Neck Neoplasms
Keywords: cancer; squamous cell; carcinoma; head; neck
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms; Carcinoma | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gefitinib (Experimental): Patients were started on gefitinib 250 mg orally daily for 2 weeks. At 2 weeks, patients were reevaluated and given skin toxicity grade according to the National Cancer Institute Common Toxicity Criteria version 3.0 (CTC 3.0). Patients with grade 2 or greater skin toxicity remained on 250 mg daily; in patients with grade 0-1 skin toxicity the dose 250-mg oral dose-escalating dose; each patient received treatment at the dose that produced grade 2 skin toxicity until disease progression or withdrawal.
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — Patients were started on gefitinib 250 mg orally daily for 2 weeks. At 2 weeks, patients were reevaluated and given skin toxicity grade according to the National Cancer Institute Common Toxicity Criteria version 3.0 (CTC 3.0). Patients with grade 2 or greater skin toxicity remained on 250 mg daily; in patients with grade 0-1 skin toxicity the dose 250-mg oral dose-escalating dose; each patient received treatment at the dose that produced grade 2 skin toxicity until disease progression or withdrawal.
  Other Names: IRESSA®

SUMMARY:
The purpose of this study is to demonstrate the activity (response rate and rate of stable disease) of Iressa administered as a single agent escalated to a dose that produces grade 2 skin toxicity in patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck (SCCHN).

DETAILED DESCRIPTION:
This open-label, multi-institution, phase II study evaluated the activity of gefitinib at individually escalated doses up to 750mg to achieve the skin toxicity grade greater than or equal to 2. Patients were started on gefitinib 250mg orally daily for 2 weeks. At 2 weeks, patients were reevaluated and given skin toxicity grade according to the National Cancer Institute Common Toxicity Criteria version 3.0 (CTC 3.0). Patients with grade 2 or greater skin toxicity remained on 250 mg daily; in patients with grade 0-1 skin toxicity the dose was escalated to 500 mg daily and again to 750 mg daily on next evaluation until grade 2 or greater skin toxicity was developed.

The protocol was later amended because of the reported lower efficacy of the 250 mg dose and patients were then started at 500 mg per day. There was no further dose escalation beyond 750 mg per day irrespective of the response or grade of skin toxicity. Therapy was discontinued upon disease progression, unacceptable toxicity, death or patient's withdrawal of consent. Dose interruptions were used as the first approach to managing the toxicity of the patients who experienced grade 3-4 non-hematological toxicities. Gefitinib was interrupted for up to a maximum of 14 days until the toxicities dropped to grade 1 or less. Adherence to therapy was monitored using drug diaries that were collected at each physician visit and assessed against pill counts.

ELIGIBILITY:
Inclusion Criteria:

* squamous cell carcinoma of the head and neck
* Tumour site that is amenable to biopsy. Patients can refuse biopsy and still participate in the study but all patients must have disease that can be biopsied
* Aged 18 years or older
* Prior epidermal growth factor receptor (EGFR) based therapy is allowed if greater than 4 months have elapsed since last dose of that agent and study entry
* No chemotherapy or irradiation within the 28-day period preceding entry to the study.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Ability to understand and the willingness to sign a written informed consent document.
* Normal organ and marrow function

Exclusion Criteria:

* Known severe hypersensitivity to Iressa or any of the excipients of this product
* Other co-existing malignancies or malignancies diagnosed within the last 3 years with the exception of basal cell carcinoma or cervical cancer in situ
* Any unresolved chronic toxicity greater than CTC grade 2 from previous anticancer therapy (except alopecia).
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the trial
* Pregnancy or breast feeding women
* Concomitant use of phenytoin, carbamazepine, rifampicin, barbiturates, or St John's Wort
* Treatment with a non-approved or investigational drug within 30 days before Day 1 of study treatment
* Any evidence of clinically active interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-03; Primary Completion 2008-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ezra EW Cohen, MD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Northwestern University, Chicago, Illinois

REFERENCES:
- [Result] Perez CA, Song H, Raez LE, Agulnik M, Grushko TA, Dekker A, Stenson K, Blair EA, Olopade OI, Seiwert TY, Vokes EE, Cohen EE. Phase II study of gefitinib adaptive dose escalation to skin toxicity in recurrent or metastatic squamous cell carcinoma of the head and neck. Oral Oncol. 2012 Sep;48(9):887-92. doi: 10.1016/j.oraloncology.2012.03.020. Epub 2012 Apr 17. PMID 22513208

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gefitinib
Started | 44
Completed | 36
Not Completed | 8
Not completed — Death | 6
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Gefitinib
Number analyzed (Participants) | 44
Age, Customized [Number; unit: participants]
  <= 62 years | 26
  > 62 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Response (CR or PR), Stable Disease (SD), and Progressive Disease (PD) Rates
Description: The proportion of subjects that responded [complete (CR) or partial response (PR)], had stable disease (SD), or progressive disease (PD) as defined by the Response Evaluation Criteria In Solid Tumors (RECIST)
  Complete Response (CR): Disappearance of all target lesions
  Partial Response (PR): At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter (LD) since the treatment started
  Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: 8 weeks
Population: Eight patients were not assessable for response, six of them died prior to the evaluation of response. For the purpose of the analysis these patients were classified as having disease progression in response to therapy.
Measure: Number; unit: percentage of participants
Arm/Group | Gefitinib
Number analyzed (Participants) | 44
percentage of participants
  Response (CR or PR) | 6.81
  Stable disease (SD) | 18.18
  Progressive disease (PD) | 75.00

2. Secondary Outcome: Median Progression-free Survival Time
Description: Progression-free survival (PFS) is the number of months during and after Gefitinib treatment during which the cancer did not get worse (progress) as defined by Response Evaluation Criteria In Solid Tumors (RECIST). Progressive disease is associated with at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. All patients developed progressive disease or died during the 9-month observation period.
Time Frame: 9 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gefitinib
Number analyzed (Participants) | 44
months | 1.9 [1.6 to 2.2]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during the 9-month observation period (including treatment phase and follow-up).
Arm/Group | Gefitinib
Serious Adverse Events (participants affected / at risk) | 20/44
Other Adverse Events (participants affected / at risk) | 17/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gefitinib (N=44)
Acute renal failure (Renal and urinary disorders) | 1 — Acute kidney failure is the rapid loss the kidneys' ability to remove waste and help balance fluids and electrolytes in the body.
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 — "Aspiration pneumonia isbronchopneumonia that develops due to the entrance of foreign materials into the bronchial tree,[1] usually oral or gastric contents (including food, saliva, or nasal secretions). "
Atrial fibrillation (Cardiac disorders) | 2 — "Atrial fibrillation is an irregular and often rapid heart rate that commonly causes poor blood flow to the body. During atrial fibrillation, the heart's atria beat chaotically and irregularly, out of coordination with the ventricles of the heart"
Bleeding from tumor site (General disorders) | 1 — Bleeding from tumor site
Bleeding from unspecified region (General disorders) | 2 — Bleeding from unspecified region
Dehydration (Gastrointestinal disorders) | 1 — "Dehydration (hypohydration) is the excessive loss of body water, with an accompanying disruption of metabolic processes."
Diarrhea (Gastrointestinal disorders) | 1 — Diarrhea is the condition of having three or more loose or liquid bowel movements per day.
Dysphagia (Gastrointestinal disorders) | 1 — Dysphagia is the medical term for the symptom of difficulty in swallowing.
Fever (General disorders) | 1 — Fever is characterized by an elevation of body temperature above the normal range of 36.5-37.5 degrees C (97.7-99.5 degrees F) due to an increase in the temperature regulatory set-point.
G-tube malfunction (General disorders) | 1 — A gastrostomy tube (also called a G-tube) is a tube inserted through the abdomen that delivers nutrition directly to the stomach. One patient was hospitalized because the G-tube stopped working properly.
G-tube placement (General disorders) | 2 — A gastrostomy tube (also called a G-tube) is a tube inserted through the abdomen that delivers nutrition directly to the stomach. Two patients were hospitalized because their gastrointestinal function declined and warranted G-tube placement.
GI bleeding (Gastrointestinal disorders) | 1 — Gastrointestinal (GI) bleeding refers to any bleeding that starts in the gastrointestinal tract.
Headache (General disorders) | 1 — A headache or cephalalgia is pain anywhere in the region of the head or neck.
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 — "Hypoxia, or hypoxiation, is apathological condition in which the body as a whole (generalized hypoxia) or a region of the body (tissue hypoxia, or less commonly regional hypoxia) is deprived of adequate oxygen supply. "
Nausea (Gastrointestinal disorders) | 2 — Nausea is a sensation of unease and discomfort in the upper stomach with an involuntary urge to vomit.
Neck bleeding (General disorders) | 1 — Bleeding from neck region
Pain (General disorders) | 1 — Patient experienced pain at grades 4 or higher.
Pericardial effusion (Cardiac disorders) | 1 — "Pericardial effusion (""fluid around the heart"") is an abnormal accumulation of fluid in the pericardial cavity."
Pleurodesis (Respiratory, thoracic and mediastinal disorders) | 1 — Pleurodesis is a procedure used to cause the layers of the lung lining (the pleura) to stick together.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 — Pneumonia is an inflammatorycondition of the lungaffecting primarily the microscopic air sacs known as alveoli.
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 — "Respiratory distress is a medical term that refers to both difficulty in breathing, and to the psychological experience associated with such difficulty, even if there is no physiological basis for experiencing such distress."
Retroperitoneal bleed (General disorders) | 1 — "Bleeding in the retroperitoneal space (retroperitoneum), i.e. the anatomical space in the abdominal cavity behind (retro) the peritoneum."
Sepsis (Infections and infestations) | 2 — Sepsis is a potentially deadly medical condition characterized by a whole-body inflammatory state (called a systemic inflammatory response syndrome or SIRS) caused by severe infection.
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 — Stridor is a high-pitched wheezing sound resulting fromturbulent air flow in the upper airway.
Subacute hemorrhage of thalamus (General disorders) | 1 — Subacute (between chronic and acute) hemorrhagic bleeding into the thalamus
Tracheitis (Respiratory, thoracic and mediastinal disorders) | 1 — Bacterial tracheitis is a bacterial infection of the trachea and is capable of producing airway obstruction.
Unresponsiveness (General disorders) | 1 — Poor response or total loss of response to questions or other stimuli
Urinary tract infection (Renal and urinary disorders) | 1 — A urinary tract infection (UTI) (also known as acute cystitis or bladder infection) is an infection that affects part of the urinary tract.
Vomiting (Gastrointestinal disorders) | 1 — Vomiting (known medically as emesis and informally as throwing up and numerous other terms) is the forceful expulsion of the contents of one's stomach through the mouth and sometimes the nose.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gefitinib (N=44)
Dehydration (Gastrointestinal disorders) | 3 — "Dehydration (hypohydration) is the excessive loss of body water, with an accompanying disruption of metabolic processes."
Dysphagia (Gastrointestinal disorders) | 4 — Dysphagia is the medical term for the symptom of difficulty in swallowing.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 — Shortness of breath
Epistaxis (Blood and lymphatic system disorders) | 3 — Nosebleed
Fatigue (General disorders) | 3 — "Fatigue (also called exhaustion, tiredness, lethargy, languidness, languor, lassitude, and listlessness) is a subjective feeling of tiredness which is distinct from weakness, and has a gradual onset."
Rash (Skin and subcutaneous tissue disorders) | 7
Xerostomia (Gastrointestinal disorders) | 3 — Xerostomia is the medical term for the subjective symptom of dryness in the mouth.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes